CLINICAL TRIAL: NCT05870670
Title: Investigation of Pharmacokinetics, Safety, and Tolerability of Multiple Subcutaneous Doses of NNC0519-0130 in Japanese and Non-Japanese Male Participants
Brief Title: A Research Study of a New Medicine NNC0519-0130 in Japanese and Non-Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9541-4921; U1111-1283-0710 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0519-0130 (Experimental): Escalating multiple doses of NNC0519-0130 administered subcutaneously.
  Interventions: Drug: NNC0519-0130
- Placebo (Placebo Comparator): Escalating multiple doses of NNC0519-0130 matching placebo administered subcutaneously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0519-0130 — Administered subcutaneously.
  Arms: NNC0519-0130
Drug: Placebo — Administered subcutaneously.
  Arms: Placebo

SUMMARY:
NNC0519-0130 is a new medicine which may possibly help participants with type 2 diabetes. This study, will look into how safe the new medicine NNC0519-0130 is, and we will measure its concentrations in the blood and look at its effects. This study will last for a maximum of 22 weeks and Japanese and Non-Japanese male participants will be included.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 23.0 kilogram per meter square (kg/m^2) and 39.9 kg/m^2 (both inclusive) at screening with a minimum weight of 50 kilogram (kg). Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* For Japanese participants: Both parents of Japanese descent.
* For non-Japanese participants: Both parents of Caucasian descent.

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions.
* Glycosylated haemglobin (HbA1c) greater than or equal to 6.5 percent (48 millimoles per mole [mmol/mol]) at screening.
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, occasional use of paracetamol, ibuprofen, acetylsalicylic acid (ASA), and domperidon, or topical medication not reaching systemic circulation, within 14 days before screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,0130, SS: Area Under the NNC0519-0130 Plasma Concentration-Time Curve After the Last Dose in Each Treatment Period | From pre-dose until 24 hours post-dose relative to last dose in each treatment period
  Measured in h*nmol/L.

SECONDARY OUTCOMES:
Cmax,0130, SS: Maximum Plasma Concentration of NNC0519- 0130 After the Last Dose in Each Treatment Period | From pre-dose until 24 hours post-dose relative to last dose in each treatment period
  Measured in nmol/L.
Number of Treatment Emergent Adverse Events (TEAEs) | From time of dosing (day 1) until completion of the follow-up visit (day 105)
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com